CLINICAL TRIAL: NCT01497210
Title: A Prospective, Multi-centre, Non-comparative Study to Evaluate the Safety and Preliminary Performance of the EASH Dressing on Chronic Venous Leg Ulcers
Brief Title: EASH Dressing on Chronic Venous Leg Ulcers
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: ConvaTec Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CW-0205-11-U356
Record Dates: First submitted 2011-12-20; First posted 2011-12-22 (Estimated); Last update posted 2012-04-25 (Estimated); Status verified 2012-04

CONDITIONS: Leg Ulcer
MeSH Terms: conditions — Leg Ulcer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- EASH (Experimental)
  Interventions: Device: EASH dressing

INTERVENTIONS:
Device: EASH dressing — Apply study dressing for 4 weeks changing at least every 7 days followed by Aquacel for four weeks.

SUMMARY:
The primary objective of this study is to evaluate the safety and preliminary performance of EASH dressing for 4 weeks followed by AQUACEL® dressing for 4 weeks on venous leg ulcers.

ELIGIBILITY:
Inclusion Criteria:

* Subjects over 18 years, willing and able to provide written informed consent.
* Subjects who have an ankle to brachial pressure index (ABPI) of 0.8 or greater
* Subjects who have a venous leg ulcer (i.e. CEAP classification of C6 1), with duration less than 24 months and size ranging between 5 cm2-40 cm2.
* Subjects' leg ulcers will meet at least 3 of the 5 following clinical signs of infection: pain between two dressing changes, peri-ulcer skin erythema/inflammation, oedema, malodour (foul odour), and heavy exudate.
* Subjects who agree to wear compression therapy daily in combination with the trial dressing.

Exclusion Criteria:

* Subjects with a history of skin sensitivity to any of the components of the study product.
* Subjects who have had current local or systemic antibiotics in the week prior to inclusion with the exception of wounds that are considered to be clinically infected at baseline.
* Subjects whose leg ulcers are malignant, or who have had recent deep venous thrombosis or venous surgery within the last 3 months.
* Subjects who have progressive neoplastic lesion treated by radiotherapy or chemotherapy, or on-going treatment with immunosuppressive agents
* Subjects exhibiting any other medical condition which, according to the Investigator, justifies the subject's exclusion from the study
* Subjects who have participated in a clinical study within the past month.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2011-11; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Safety | All 8 weeks
  Nature and frequency of adverse events.

SECONDARY OUTCOMES:
Ulcer Improvement (wound bed) | Baseline, week 4 and week 8
Ulcer Improvement (peri-ulcer) | Baseline, week 4 and week 8 or final visit
Healing | Weekly for 4 weeks then biweekly for 4 weeks or final visit
  Reduction in ulcer area
Healing | 8 weeks or final visit
  Number of subjects healed
Healing | 8 weeks or final visit
  Time to healing
Ulcer pain | Weekly for 4 weeks then biweekly for 4 weeks or final visit
Comfort | Weekly for 4 weeks then biweekly for 4 weeks
Ease of use | Weekly for 4 weeks then biweekly for 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Keith Harding, Principal Investigator — Wound Healing Research Unit, Cardiff University
Locations (6):
- Poland (3):
  - Mikomed, Lodz
  - Cross Medica, Warsaw
  - Medservice, Zabrze
- United Kingdom (3):
  - Wound Healing Research Unit, Heathpark, Cardiff
  - Axbridge & Wedmore Medical Practice, Axbridge, Somerset
  - Arrowe Park Hospital, Upton, Wirral